CLINICAL TRIAL: NCT04134962
Title: Evaluation of a New Tool for Measuring Hindfoot Alignment Under Load and in 3D. 3D-HAM Study.
Brief Title: Evaluation of a New Tool for Measuring Hindfoot Alignment Under Load and in 3D.
Acronym: 3D-HAM
Status: Completed | Type: Observational
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr François Lintz (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-A01178-45
Record Dates: First submitted 2019-10-03; First posted 2019-10-22 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Ankle Surgery; Foot Surgery; 3D Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ankel surgery group: Adult patients for which a Cone Beam under load is prescribed for a preoperative assessment of a foot or ankle surgery or for a follow-up consultation.
  Interventions: Diagnostic Test: 3D Imaging FAO measurement and Clinical evaluation of the hindfoot alignment
- control foot group: Adult patients for which a Cone Beam under load is prescribed for a preoperative assessment of a foot or ankle surgery or for a follow-up consultation.
  Will be retained only results of normal aligment FAO
  Interventions: Diagnostic Test: 3D Imaging FAO measurement and Clinical evaluation of the hindfoot alignment

INTERVENTIONS:
Diagnostic Test: 3D Imaging FAO measurement and Clinical evaluation of the hindfoot alignment — The Cone Beam under load is used for the diagnosis and monitoring of the foot and ankle. It has a CE marking for this purpose.
  The images obtained by the Cone Beam under load (Ped Cat) will be analysed using the TALAS mathematical algorithm tool to measure the FAO.
  The internal software of the Cone Beam under load will also be used to obtain a "radiographic" image corresponding to a 2D projection on which the tibio-calcaneal angle can be measured.

SUMMARY:
The automated TALAS measurement tool, working with the Cone Beam 3D scanner under load, provides a reproducible measurement of the Foot Ankle Offset (FAO). It is possible to determine an average value and the standard deviation of FAO in the relevant population. And to differentiate significantly the populations with a neutral alignment, varus or valgus.

DETAILED DESCRIPTION:
The analysis of the alignment of the foot is fundamental in the management of pathologies of the foot and ankle. The advent of 3D imaging under load (Scanner Cone Beam), less radiant and more precise, requires the development and evaluation of new measurement tools.

The automated TALAS measurement tool, working with the Cone Beam 3D scanner under load, provides a reproducible measurement of the Foot Ankle Offset (FAO). It is possible to determine an average value and the standard deviation of FAO in the relevant population. And to differentiate significantly the populations with a neutral alignment, varus or valgus.

ELIGIBILITY:
Inclusion Criteria:

* Patient selected for a preoperative assessment in foot or ankle surgery, or patient seen in follow-up consultation for which a Cone Beam under load is prescribed
* Patient having been informed of this study and having given their consent
* Patient over 18 years old
* Unprotected adult

Exclusion Criteria:

* Patient with a contraindication to the Cone Beam under load
* Patient refusing to participate in this study
* Non-plantigrade foot under load (impossibility of simultaneously resting M1, M5 and Calcaneus on the ground)
* Patient who has already participated in the 3D HAM study (patients who would have participated in the study during the preoperative consultation for which another Cone Beam would be prescribed during the follow-up consultation. These patients would not be able to participate again in this study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult's patients for which a Cone Beam under load is prescribed for a preoperative assessment of a foot or ankle surgery or for a follow-up consultation.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
FAO value measured | 1 day
  - FAO value measured using the TALAS tool on data collected by the Cone Beam under load (PedCat). For the descriptive study of the distribution within the different populations (varus/normal/valgus), the first measurement carried out will be represented.
FAO Reliability | 1 day
  - reliability of FAO measurement by the TALAS tools (Intraclass correlation coefficient)
FAO sensitivity-specificiy | 1 day
  - Couples (Sensitivity - Specificity) of the FAO ROC curve allowing the morphological classification of the patients (Varus, Valgus or Normal)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de L'Union, Saint-Jean, France

IPD SHARING:
Plan to Share IPD: Undecided